CLINICAL TRIAL: NCT00997555
Title: Prophylactic Bronchoscopy After Inhalation Injury in Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hurley Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMC0001
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Results first posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2012-12

CONDITIONS: Inhalation Injury; Pneumonitis; Pneumonia
Keywords: inhalation; bronchoscopy; burn; pneumonia
MeSH Terms: conditions — Pneumonia; Respiratory Aspiration; Burns | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bronchoscopy intervention group (Experimental): Group undergoing scheduled bronchoscopy.
  Interventions: Procedure: bronchoscopy
- Control group (No Intervention): Standard treatment without scheduled bronchoscopy.

INTERVENTIONS:
Procedure: bronchoscopy — Scheduled bronchoscopy.
  Arms: bronchoscopy intervention group

SUMMARY:
The investigators hypothesize that the scheduled use of bronchoscopy on a regular basis after inhalation injury in burn patients will improve outcome by providing pulmonary hygiene, decrease the incidence of pneumonia, and detect pneumonia earlier than standard treatment without bronchoscopy.

DETAILED DESCRIPTION:
The role of bronchoscopy in most hospitals has been limited to obtaining lavage fluid for culture and assessing the degree of airway injury, which has been shown to be predictive of outcome. Severe inhalation injury, which is characterized by pulmonary edema, bronchial edema, and secretions, can occlude the airway and lead to atelectasis and pneumonia. Aggressive use of bronchoscopy is highly effective in removing foreign particles and accumulated secretions that worsen the inflammatory response and impede ventilation. While it seems intuitive that bronchoscopy would improve pulmonary hygiene by removing secretions and denuded epithelial slough in burn patients, there has not been any published data to support or deter the use of bronchoscopy for inhalation injury nor document an improvement in morbidity or mortality secondary to bronchoscopy as a therapeutic intervention.

Recent research has shown that the process of intubation for mechanical ventilation provides a portal for bacterial contamination, after which the damaged tracheobronchial mucosa quickly becomes colonized with pathogenic organisms in over 50% of the patients. Furthermore, within 15 minutes of smoke inhalation, there is significant airway edema and thickening, more prominently in the lower trachea than the upper portion. These factors place the patient with inhalation injury at high risk for pneumonia.

We have used the National Burn Repository data to previously show that patients who receive aggressive use of bronchoscopy after inhalation injury have an improved outcome in terms of decreased ventilator days, decreased ICU length of stay, decreased incidence of pneumonia, and a trend towards improved mortality. However, that data was unable to document why. It was also unable to confirm that the findings were not due to institutional bias. Therefore, one of the conclusions from that study was that a prospective trial is needed to confirm the findings.

Our hypothesis is that a scheduled and sequential use of bronchoscopy after inhalation injury as a therapeutic tool to remove secretions, slough, carbonaceous material, and screen for the early detection of pneumonia by bronchoalveolar lavage (BAL) will improve outcome. We will attempt to document this improvement by using the following endpoints: length of ICU stay, length of hospital stay, ventilator days, incidence of pneumonia, overall morbidity and mortality with and without bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Any burned patient arriving intubated on mechanical ventilation OR requiring mechanical ventilation within 48 hours of admission AND
2. > 18 years old AND
3. patient believed to be able to survive more than 48 hours after arrival (not likely to be made DNR or comfort care) including:

   * any methamphetamine explosion or
   * any burn associated with fire (not chemical) of the face or blast injury to the face or
   * confined in a burning space for more than 10 minutes or
   * any burn with carbonaceous material around the nose or mouth or
   * any burn > 15% TBSA associated with fire (not chemical) or
   * any burn associated with an explosion in a confined space.

Exclusion Criteria:

1. Likely to die within 48 hours based upon severity of injury.
2. Less than 18 years old.
3. Burned patient transferred to our facility already on mechanical ventilation for more than 48 hours.
4. Patient already on antibiotics for another reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Carr, MD, Principal Investigator — Hurley Medical Center
Locations (1):
- Hurley Medical Center, Flint, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2009-2012, 33 patients with inhalation injury were admitted to our regional burn center.
Pre-assignment Details: Five were never enrolled. Two patient's families refused to consent, and two fell into exclusion criteria number 1. Both died within six hours of admission. The remaining fifth patient self-extubated and thus failed to meet inclusion criteria number 1. This left 28 patients for analysis, all of whom were enrolled and randomized into the study.
Groups:
- Bronchoscopy Intervention Group: Group undergoing scheduled bronchoscopy. Patients had bronchoscopy and BAL performed within 12 hours of arrival and every 3 days sequentially. A positive BAL (> 100K CFU/ml) were treated with antibiotics according to sensitivites.
Period: Overall Study
Arm/Group | Bronchoscopy Intervention Group | Control Group
Started | 13 | 15
Completed | 13 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bronchoscopy Intervention Group | Control Group | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 15 | 23
  >=65 years | 5 | 0 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (11) | 35 (8) | 42 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality
Description: Bronchoscopy group deaths n=0. Control group deaths n=1.
Time Frame: until death or discharge from hospital, data reviewed every 6 months
Measure: Number; unit: participants
Arm/Group | Bronchoscopy Intervention Group | Control Group
Number analyzed (Participants) | 13 | 15
participants | 0 | 1

2. Primary Outcome: Respiratory Associated Mortality
Description: Bronchoscopy group deaths n=0. Control group deaths n=1.
Time Frame: until death or discharge from hospital, data reviewed every 6 months
Measure: Number; unit: participants
Arm/Group | Bronchoscopy Intervention Group | Control Group
Number analyzed (Participants) | 13 | 15
participants | 0 | 1

3. Secondary Outcome: Incidence of Pneumonia
Description: Bronchoscopy group- 4/13 (31%) Control group- 6/15 (40%)
Time Frame: until discharge from the hospital, data reviewed every 6 months
Measure: Number; unit: participants
Arm/Group | Bronchoscopy Intervention Group | Control Group
Number analyzed (Participants) | 13 | 15
participants | 4 | 6
Statistical Analysis 1: Comparison: Bronchoscopy Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.6, Chi-squared

4. Secondary Outcome: Length of Mechanical Ventilation
Description: Days of mechanical ventilation (bronchoscopy 5.1 days, 95% CI +/- 3.6 days versus control 6.7 days, 95% CI +/- 6.3 days, p = 0.7).
Time Frame: until discharge from hospital, data reviewed every 6 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bronchoscopy Intervention Group | Control Group
Number analyzed (Participants) | 13 | 15
days | 5.1 [2.5 to 8.7] | 6.7 [0.4 to 13.0]
Statistical Analysis 1: Comparison: Bronchoscopy Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.7, t-test, 2 sided — (bronchoscopy 5.1 days, 95% CI +/- 3.6 days versus control 6.7 days, 95% CI +/- 6.3 days, p = 0.7)

5. Secondary Outcome: Length of ICU Stay
Description: Number of ICU days (bronchoscopy 10 days, 95% CI +/- 10 days versus control 18 days, 95% CI +/- 12 days, p = 0.4).
Time Frame: until discharge from hospital, data reviewed every 6 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bronchoscopy Intervention Group | Control Group
Number analyzed (Participants) | 13 | 15
days | 10 [0 to 20] | 18 [6 to 30]
Statistical Analysis 1: Comparison: Bronchoscopy Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.4, t-test, 2 sided; (bronchoscopy 10 days, 95% CI +/- 10 days versus control 18 days, 95% CI +/- 12 days, p = 0.4)

6. Secondary Outcome: Length of Hospital Stay
Description: Number of hospital days (bronchoscopy 21 days, 95% CI +/- 12 days versus control 26 days, 95% CI +/- 12 days, p = 0.5).
Time Frame: until discharge from hospital, data reviewed every 6 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bronchoscopy Intervention Group | Control Group
Number analyzed (Participants) | 13 | 15
days | 21 [9 to 33] | 26 [14 to 38]
Statistical Analysis 1: Comparison: Bronchoscopy Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.5, t-test, 2 sided; (bronchoscopy 21 days, 95% CI +/- 12 days versus control 26 days, 95% CI +/- 12 days, p = 0.5)

ADVERSE EVENTS:
Arm/Group | Bronchoscopy Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes